CLINICAL TRIAL: NCT04302233
Title: A Randomized, Controlled Study of the Superiority Between 2 Types of POSToperative Pharmaceutical Support on Patients' Knowledge of Their IMPlant: Breast or Joint Prostheses
Brief Title: A Randomized Study of Superiority of POSToperative Pharmaceutical Support on Patients' Knowledge of Their IMPlant
Acronym: POSTIMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP200083
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Joint Prosthesis; Breast Implants; Health Education
Keywords: joint prosthesis; breast implants; health education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicentric, controlled, single-blind, randomized trial in two parallel arms
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New pharmaceutical support (NPS) (Experimental): An NPS is an interview comprising the following elements:
  The delivery of the identification sheet of their implants with:
  * a quiz to focus the patient's attention
  * a description of the characteristics of their prosthesis using a specific photo of their implant
  * a presentation of the medical device vigilance.
  * an explanation of the value of the identification sheet for their implant, An in-depth presentation of an information booklet on living at home with their prosthesis and on medical and paramedical monitoring.
  For patients in orthopedic surgery: a booklet specific to their prosthesis and the surgical approach For plastic surgery patients, the information sheets published by the French Society of Plastic Reconstructive and Aesthetic Surgery (SOF.CPRE).
  A time to answer any questions the patient may have
  Interventions: Other: New pharmaceutical support (NPS)
- Usual pharmaceutical support (UPS) (No Intervention): An UPS is an interview comprising the following elements:
  * The delivery of the same patient-implant sheet as in arm 1, but without additional oral information.
  * The delivery and oral presentation of the same booklet as practiced in the arm 1 (NPS).
  * And a time to answer any questions from the patient months

INTERVENTIONS:
Other: New pharmaceutical support (NPS) — The only difference between these 2 groups is that patients in the NPS group benefit from additional visual and oral information on the characteristics of their implant and on medical device vigilance during their hospitalization.
  Arms: New pharmaceutical support (NPS)

SUMMARY:
Recently joint and breast prostheses were placed under special post-marketing surveillance in order to prevent new occurrence of serious incidents by agency for medicines and health products safety. Few of french patient are able to identify their prosthesis in the event on health security alert. An usual postoperative pharmaceutical support (UPS) for patients with joint prosthesis has been implemented to prepare them for return home. At the request of surgeons, a new pharmaceutical support (NPS) has been developed to improve the ability of these patients to recall or find information that identify their prosthesis.

Objectives :

The main objective is to demonstrate that the new pharmaceutical support (NPS) increase the ability to memorize then find correct information of their prosthesis 6 months post-implantation

Material and method :

This study, approved by an ethic committee, takes place in the orthopedic and plastic surgery departments. The 236 adult patients included are hospitalized following the scheduled placement of either a breast or a hip or knee prosthesis. They are randomized, either in the NPS group or in the UPS comparator group. In both cases, patients benefit from the same written information: a patient-implant file and an information booklet specific to their prosthesis, validated by specialist surgeons, to prepare for their return home. The only difference between these 2 groups is that patients in the NPS group benefit from additional visual and oral information on the characteristics of their implant and on medical device vigilance during their hospitalization. In NPS group, pharmacist use specific photo and quiz.

A telephone follow-up at the 6th month of the patients is carried out by a pharmacist to assess the patient's knowledge, using a standardized questionnaire.

Expected results :

Based on retrospective data already published, the main hypothesis is that the NPS is associated with an improvement in patient ability to remember the correct model or manufacturer of their prosthesis, compared to the UPS, 6 months after the operation.Secondary hypotheses are that NPS compared to UPS leads to an improvement in patients ability to preserve and find correct items related to theirs prosthesis at 6 months as well as an improvement in their knowledge of medical device vigilance and patient satisfaction declarations and a decrease in anxiety associated with prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient hospitalized following the scheduled placement of one of the following prostheses: three-compartment knee prostheses or total hip prosthesis or breast implant
* French-speaking or non-French-speaking patient accompanied by a French-speaking support person
* Patient having received complete information and having signed a free and informed consent for the research
* Patient affiliated to a social security scheme (beneficiary or entitled)

Exclusion Criteria:

* Patient having been operated on for the installation of an orthopedic prosthesis not programmed within the framework of a trauma emergency.
* Patient suffering from post-operative confusional syndrome;
* Non-French speaking patient unaccompanied or accompanied by a non-French speaking support person
* Patient on state medical aid
* Persons referred to in articles L1121-5, 6 and 8 of the public health code (corresponds to protected persons): pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to legal protection measure, hospitalized for psychiatric disorder.
* Patient who has already had postoperative pharmaceutical support for the placement of the same type of prosthesis on the contralateral limb
* Patient suffering from a known cognitive or memory disorder.
* Patient expressly refusing to participate in the telephone interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
pourcentage of patients able to recall the correct name of the manufacturer brand or model of their prosthesis after traceability checking by a questionnaire at 6 months postoperative. | 6 month

SECONDARY OUTCOMES:
pourcentage of patients who recall the reception of a patient-implant file during hospitalization by a questionnaire at 6 months postoperative. | 6 month
pourcentage of patients able to identify three correct information after traceability checking on the implantation, by a questionnaire at 6 months postoperative | 6 month
  The three requested information are on the card or patient-implant sheet for this outcome are following :
  Item 1 : Accurate date of implantation : Date as DD/MM/YYYY format Item 2 : Surgeon's name who placed their prosthesis Item 3 : Batch number of one of the DMI composing their prosthesis : For hip prosthesis, question is about femoral head and for knee prosthesis, question is about tibial insert. If there is implantation of 2 breast prostheses, this is data from right prosthesis which are requested.
pourcentage of patients who recall health institution where the prosthesis was implanted by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients who know there is a regular medical monitoring after implantation by a questionnaire at 6 months postoperative. | 6 month
pourcentage of patients who recall material (s) composing the prosthesis by a questionnaire at 6 months postoperative. | 6 month
  Ability of patients to recall correct and useful characteristics for the identification of their prosthesis in the event of a descending health alert (so that the patient knows if he is affected by this alert)
pourcentage of patients with breast implants who recall shape (anatomical or round) and surface texturing (smooth or textured) after traceability checking by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients with hip prosthesis who recall the location of the operative scar (anterior or posterolateral) and fixing method of the prosthesis (with ciment or without) by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients know they can report an adverse effect associated with the prosthesis by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients know institutions able to receive an adverse effect associated with the prosthesis (French agency for medicines and health products (ANSM), industrial, surgeon, other) by a questionnaire at 6 months postoperative. | 6 month
pourcentage of patients know a prosthesis traceability document (Hospital report, patient card and patient sheet) by a questionnaire at 6 months postoperative. | 6 month
pourcentage of patients having called the care service and average of call by patient by a questionnaire at 6 months postoperative. | 6 month
  This outcome is an association of four items to assessed the quality and quality medical needs after implantation
pourcentage of patients having consulted outside of Mondor hospital and average of consultation by patient by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients have been admitted to the emergency by a questionnaire at 6 months postoperative. | 6 month
pourcentage of patients have been admitted to the hospitalization for a complication related to the prosthesis by a questionnaire at 6 months postoperative | 6 month
pourcentage of patients having worn already at least one prosthesis before the day of intervention by a questionnaire. | 6 month
pourcentage of patients wearing always a prosthesis among patient wearing already prostheses keep prosthesis before the day of intervention by a questionnaire. | 6 month
Average of implant / prosthesis by patient before the day of intervention by a questionnaire. | 6 month
pourcentage of patients having already a hip, a knee, a breast or an active implantable medical device implant before the day of intervention by a questionnaire | 6 month
pourcentage of patients knowing all or someone or no one manufacturer name or model of each prosthesis in place before the day of intervention by a questionnaire. | 6 month
pourcentage of patients knowing the implantation year of each prosthesis before the day of intervention by a questionnaire. | 6 month
pourcentage of patients able to give the health institution name where previous implant(s) were placed by a questionnaire (Mondor hospital or others). | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: Yes
data are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information